CLINICAL TRIAL: NCT05597176
Title: Telemonitored Exercise to Attenuate Metabolic Dysregulation in Spinal Cord Injury (TEAM-SCI)
Brief Title: Telemonitored Exercise to Attenuate Metabolic Dysregulation in Spinal Cord Injury
Acronym: TEAM-SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Eduard Tiozzo, PhD, Research Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220652
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Spinal Injuries
MeSH Terms: conditions — Spinal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal Cord Injury Exercise Group (Experimental): Participants will exercise at home 3-5 times per week under supervision via teleconference. Participants will be part of this group for 18-20 weeks.
  Interventions: Other: Spinal Cord Injury Exercise Group

INTERVENTIONS:
Other: Spinal Cord Injury Exercise Group — Participants will have an initial accommodation period of 4 weeks, during which four 10-minute exercise bouts/day will be interspersed with 5 minutes of rest. The bouts will gradually increase until at least continuous 40-minute sessions. The remaining 12-week intervention will be set at 70% max heart rate for a total of 16 weeks.

SUMMARY:
The purpose of this research is to test the health benefits of using functional electrical stimulation for lower extremity exercise at home.

DETAILED DESCRIPTION:
The specific objectives are to assess the impact of 16 weeks of home-based telemonitored functional electrical stimulation leg cycle ergometry (FESLCE) exercise on body composition and metabolic health in adults with C4-T4 motor complete SCI. This study is available only to those who were previously enrolled in the SCIENCE protocol #20190659 that were randomized to the diet alone group. After completing the dietary intervention, those individuals will have an opportunity to experience FES bicycle.

ELIGIBILITY:
Inclusion Criteria:

* Women of child-bearing potential who agree to refrain from getting pregnant during the trial
* Previously enrolled in the SCIENCE protocol (NCT03495986) randomized to the diet alone group in SCIENCE, and are willing to complete an 8-week (2 month) washout period after the completion of the dietary intervention in the study.

Exclusion Criteria:

* Do not meet inclusion criteria above
* Those who have participated in a Functional Electrical Stimulation (FES) or ACE exercise program (>60 minutes/week) within the past 3 months
* Self-reported or documented history of:

  * orthopedic limitations
  * coronary artery disease
  * type 1 diabetes mellitus; insulin-requiring Type 2 diabetes mellitus; untreated Type 2 diabetes mellitus
  * untreated hypothyroidism
  * renal disease
  * uncontrolled autonomic dysreflexia, recent (within 3 months)
  * deep vein thrombosis (within the past 3 months)
* On anticoagulation therapy
* Pressure injuries > Grade II
* Decisional impairment
* Prisoners
* Pregnant or nursing women
* Any potential causes of autonomic dysreflexia at the discretion of the PI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Change in percent body fat | Baseline, 20 weeks (Post Intervention)
  Percent body fat will be assessed using Dual Energy x-ray absorbency (DXA)
Change in percent visceral fat | Baseline, 20 weeks (Post Intervention)
  Percent visceral fat will be assessed using DXA
Change in percent of lean body mass | Baseline, 20 weeks (Post Intervention)
  Percent lean body mass will be assessed using DXA
Change in percent of fat free mass | Baseline, 20 weeks (Post Intervention)
  Percent fat free mass will be assessed using DXA

SECONDARY OUTCOMES:
Change in Lipid Panel values | Baseline, 20 weeks (Post Intervention)
  Lipid panel values including High Density Lipoprotein, Low Density Lipoprotein, Total Cholesterol and triglycerides, all assessed in mg/dL, will be measured from blood samples
Change in resting metabolic rate | Baseline, 20 weeks (Post Intervention)
  Change in resting metabolic rate will be measured by using a large clear plastic dome over the head and the air exhaled will be measured
Change in glucose levels | Baseline, 20 weeks (Post Intervention)
  Glucose will be measured in mg/dL using blood samples
Change in HgbA1C levels | Baseline, 20 weeks (Post Intervention)
  Hemoglobin A1c (HgbA1c) levels will be assessed using blood samples
Change in Insulin levels | Baseline, 20 weeks (Post Intervention)
  Insulin levels will be assessed using blood samples
Change in hsCRP levels | Baseline, 20 weeks (Post Intervention)
  High sensitivity C Reactive Protein (hsCRP) will be assessed using blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Tiozzo, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Christine E. Lynn Rehabilitation Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No